CLINICAL TRIAL: NCT02527096
Title: A Pilot Trial Evaluating Maintenance Therapy With Lamivudine(Epivir®) and Dolutegravir(Tivicay®) in Human Immunodeficiency Virus 1 (HIV-1) Infected Patients Virologically Suppressed With Triple HAART - ANRS 167 Lamidol
Brief Title: A Trial Evaluating Maintenance Therapy With Lamivudine (Epivir®) and Dolutegravir (Tivicay®) in Human Immunodeficiency Virus 1 (HIV-1) Infected Patients Virologically Suppressed With Triple Highly Active Antiretroviral Therapy (HAART) (ANRS 167 Lamidol)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 167 Lamidol; 2015-001492-44 (EudraCT Number)
Record Dates: First submitted 2015-08-06; First posted 2015-08-18 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: HIV-1 Infection
Keywords: dolutegravir(Tivicay®); lamivudine(Epivir®); HIV-1; efficacy; safety
MeSH Terms: interventions — dolutegravir; Clinical Trials, Phase I as Topic; Lamivudine; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dolutegravir(Tivicay®) and lamivudine(Epivir®) (Experimental)
  Interventions: Drug: dolutegravir (Tivicay®) - Phase 1; Drug: lamivudine (Epivir®) - Phase 2; Drug: dolutegravir (Tivicay®) - Phase 2

INTERVENTIONS:
Drug: dolutegravir (Tivicay®) - Phase 1 — • Phase 1 (8 weeks) : switch of the third agent with dolutegravir(Tivicay®) 50 mg once a day.
Drug: lamivudine (Epivir®) - Phase 2 — • Phase 2 (48 weeks): combination with lamivudine (Epivir®) 300 mg once a day + dolutegravir (Tivicay®) 50 mg once a day. Only participants with plasma HIV RNA ≤ 50 cp/mL at Week 8 will continue on phase 2.
Drug: dolutegravir (Tivicay®) - Phase 2 — • Phase 2 (48 weeks): combination with lamivudine (Epivir®) 300 mg once a day + dolutegravir (Tivicay®) 50 mg once a day. Only participants with plasma HIV RNA ≤ 50 cp/mL at Week 8 will continue on phase 2.

SUMMARY:
The principal objective is to evaluate the antiviral efficacy of 48 weeks treatment with the two-drugs combination dolutegravir(Tivicay®) and lamivudine(TEpivir®) in HIV-1 infected patients virologically suppressed with triple HAART.

DETAILED DESCRIPTION:
Secondary objectives:

The following parameters will be evaluated :

* Evolution of CD4 cells and CD8 cells
* Tolerance to treatment
* Emergence of resistance mutations at time of virological failure
* HIV viral load measured with ultrasensitive assay (threshold 1 copy/mL) at Day 0, Week 8, Week 32 and Week 56
* Influence of total DNA at Day 0 on the occurrence of virological failure or blip
* Plasma levels of dolutegravir(Tivicay®) and lamivudine in participants with virological failure
* Adherence to treatment
* Quality of life
* Medico-economic aspects
* Dolutegravir(Tivicay®) and Nucleosidic Reverse Transcriptase Inhibitors (NRTIs) levels, and HIV viral load in semen in a subgroup of 20 participants.

Methodology:

Pilot trial, multicentric, national, prospective, no randomized and no comparative.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patient
* Age ≥ 18 years
* CD4 cell count nadir > 200/mm3
* Genotype on pre-HAART interpreted with the last version of the ANRS AC11 resistance group's algorithm which presents:

  * no major mutation on protease among: D30N, V32I, M46I/L, I47A/V, G48V, I50L/V, 154M/L, L76V, V82A/F/T/S, I84V, N88D/S, L90M,- no mutation on RT (except the mutation A98S if the patient is not infected by the virus subtype C),
  * no mutation on integrase (if the genotype is available),
* First-line treatment with suppressive triple HAART (2 NRTI + either 1 PI/r, 1 NNRTI or 1 INI). The initial treatment may have changed a maximum of two times but only once for toxicity (changes such Epivir / Ziagen to Kivexa, are not considered as a change of treatment). However, treatment has to be unchanged in the last 6 months
* Plasma HIV RNA ≤ 50 copies/mL for ≥ 2 years with at least 2 viral load determinations per year. Blips (HIV viral load between 50 and 200 copies/mL but ≤ 50 copies/mL on control sample) are allowed except in the last 6 months. The total number of blips must not exceed 3 in the last 2 years
* Negative Hepatitis Bs Antigen
* Effective contraception for women of childbearing potential
* Informed consent form signed by patient and investigator
* Patient enrolled in or a beneficiary of a Social Security programme (State Medical Aid ("Aide Médicale d'Etat" AME in France) is not a Social Security programme)

Exclusion Criteria:

* HIV-2 infection
* Positive HBc Ac isolated
* Hepatitis B Virus (HBV) co-infected patients (positive Hepatitis Bs Ag at inclusion)
* Chronic hepatitis C currently treated or needing therapy in the next 12 months
* History of HIV-associated neurocognitive disorders
* Current pregnancy or breastfeeding
* No effective contraception for the women of childbearing
* Previous treatment with chemotherapy (except bleomycin on Kaposi disease's treatment) or immunotherapy
* Grade > 2 abnormality for usual biological parameters (liver function tests, blood cell count)
* ALT(Alanine Aminotransferase) ≥ 5 x upper limit of normal value (ULN) or AST (Aspartate Aminotransferase) ≥ 3 x ULN and bilirubinemia ≥ 1.5 x ULN (with 35% direct bilirubinemia)
* Unstable liver disease (ascitis, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal or gastric varices or persistent jaundice)
* Known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Creatininemia clearance below 50 mL/min (Cockroft-Gault method)
* History or presence of allergy to the trial drugs or their components
* Severe hepatic insufficiency (Child Pugh Class C)
* Patients participating in another clinical trial including an exclusion period that is still in force during the screening phase
* Patients under "sauvegarde de justice" (judicial protection due to temporarily and slightly diminished mental or physical faculties) or under legal guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Virological success without any intercurrent event leading to interrupt the strategy of the trial (analysis) | from week 8 to week 56 (± 4 weeks)
  Virological failure is defined by plasma HIV RNA > 50 cp/mL on 2 following samples at 2 to 4 weeks apart.

SECONDARY OUTCOMES:
Evolution of CD4 and CD8 lymphocytes count (analysis) | from week 8 to week 32 and week 56
  Evaluation was calculated as the CD4 count at the corresponding week minus the baseline CD4 count
Percentage of participants who discontinued the strategy of the trial for toxicity or with adverse event of grade 3 or 4 (analysis) | week 56
Profile of resistance mutations in plasma in case of virological failure | week 56
Percentage of participants with plasma HIV RNA < 1 cp/mL | Day 0, week 8, week 32 and week 56
Influence of total DNA on the occurrence of virological failure or blip | from Day 0 to week 56
  Influence of total DNA at Day 0 on the occurrence of virological failure or blip
Measure of concentrations of dolutegravir(Tivicay®) and lamivudine(Epivir®) in case of virological failure or with a blip | week 56
Measure of adherence to treatment (self-reported) | Day 0, week 4, week 8, week 32 and week 56
Measure of quality of life (self-reported) | Day 0, week 8 and week 56
Comparison of Medico-economic substudy (analysis) | week 56
  Evaluation of medico-economic aspects. Evaluate the direct medical cost related to dolutegravir and lamivudine versus the cost of the previous treatment.
Sperm substudy measure of concentration | Week 8 and week 32
  Measure of concentrations of dolutegravir and NRTI, and HIV RNA in semen at Week 8 and Week 32 in a subgroup of 20 participants

CONTACTS AND LOCATIONS:
Overall Officials: Véronique JOLY, MD, Principal Investigator — Service des Maladies Infectieuses, Hôpital Bichat-Claude Bernard, Paris; Yazdan YAZDANPANAH, MD, Study Chair — Service des Maladies Infectieuses, Hôpital Bichat-Claude Bernard; Roland LANDMAN, MD, Study Director — Institut de Médecine et Epidémiologie Appliquée (IMEA), Paris
Locations (18):
- France (18):
  - Hôpital Avicenne, Bobigny
  - Hôpital Saint-André, Bordeaux
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital du Bocage, Dijon
  - Hôpital Pierre Zobda-Quitman, Fort de France
  - Hôpial Bicêtre, Le Kremelin Bicêtre
  - Hôpital Gui de Chaudiac, Montpellier
  - Hôpital de l'Hotel Dieu, Nantes
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Necker, Paris
  - Hôpital Bichat, Paris
  - Centre hospitalier de Pernignan, Perpignan
  - Hôpital Pontchaillou, Rennes
  - Hôpital Purpan, Toulouse
  - Hôpital Gustave Dron, Tourcoing
  - Hôpital Bretonneau, Tours

REFERENCES:
- See also: Related Info — http://www.anrs.fr/